CLINICAL TRIAL: NCT02253017
Title: Assessment Practices Registry in Congenital Cataract Surgery and Infantile
Brief Title: Evaluation of Therapeutic Strategies in Pediatric Cataract Surgery
Acronym: EP3C
Status: Withdrawn | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-06-13
Record Dates: First submitted 2014-09-26; First posted 2014-10-01 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Cataract
Keywords: Therapeutic strategies; Pediatrics; Cataract; Surgery; Intra-ocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children operated on for cataract
  Interventions: Other: Children operated on for cataract

INTERVENTIONS:
Other: Children operated on for cataract — Compilation of results of monitoring of children aged 8 to 10 months, 3 years, 5 years, 8 years

SUMMARY:
The purpose of this observational study is to assess the therapeutic strategies in the treatment of pediatric cataracts.

DETAILED DESCRIPTION:
Technical progress and recently described potential issues have recently challenged the surgical treatment of pediatric cataracts. Many questions remain unsolved: primary vs secondary implantation, nature of the implant used. The aim of this study is to establish a systematic prospective register of all cataracts operated on in a tertiary pediatric centre in order to help answering these questions.

ELIGIBILITY:
Inclusion Criteria:

* Child cataract surgery from 1 September 2014 in the Department of Ophthalmology, University Hospital Necker-Enfants Malades
* Children aged between 0 and 17 years
* Child with unilateral or bilateral cataract

Exclusion Criteria:

* Child with bilateral cataract, one eye having previously been operated in another center.
* Children whose parents have notified the doctor their refusal of data collection

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ophthalmology department, Necker hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09 (Estimated); Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment practices in Pediatric Cataract Surgery. | 8-10 months,
  * Rating of efficacy of surgery depending on the implementation or not of a primary location
  * Evaluate the effectiveness of the implementation based on the type of implant (monofocal or multifocal)
  * Evaluation of effectiveness of surgery based on age (<8 weeks of age for unilateral surgery and <11 weeks of life for bilateral surgeries)
  * To assess the frequency of adverse events, particularly glaucoma depending on the occurrence or non-implementation of a primary
Assessment practices in Pediatric Cataract Surgery. | 3 years
  * Rating of efficacy of surgery depending on the implementation or not of a primary location
  * Evaluate the effectiveness of the implementation based on the type of implant (monofocal or multifocal)
  * Evaluation of effectiveness of surgery based on age (<8 weeks of age for unilateral surgery and <11 weeks of life for bilateral surgeries)
  * To assess the frequency of adverse events, particularly glaucoma depending on the occurrence or non-implementation of a primary
Assessment practices in Pediatric Cataract Surgery. | 5 years
  * Rating of efficacy of surgery depending on the implementation or not of a primary location
  * Evaluate the effectiveness of the implementation based on the type of implant (monofocal or multifocal)
  * Evaluation of effectiveness of surgery based on age (<8 weeks of age for unilateral surgery and <11 weeks of life for bilateral surgeries)
  * To assess the frequency of adverse events, particularly glaucoma depending on the occurrence or non-implementation of a primary
Assessment practices in Pediatric Cataract Surgery. | 8 years (or 6 months after surgery if the child is carried out after 8 years )
  * Rating of efficacy of surgery depending on the implementation or not of a primary location
  * Evaluate the effectiveness of the implementation based on the type of implant (monofocal or multifocal)
  * Evaluation of effectiveness of surgery based on age (<8 weeks of age for unilateral surgery and <11 weeks of life for bilateral surgeries)
  * To assess the frequency of adverse events, particularly glaucoma depending on the occurrence or non-implementation of a primary

SECONDARY OUTCOMES:
Type of surgery and surgical procedures | 8-10 months
Type of surgery and surgical procedures | 3 years
Type of surgery and surgical procedures | 5 years
Type of surgery and surgical procedures | 8 years (or 6 months after surgery if the child is carried out after 8 years).
  8 years (or 6 months after surgery if the child is carried out after 8 years).
Type of implant | 8-10 months
Type of implant | 3 years
Type of implant | 5 years
Type of implant | 8 years (or 6 months after surgery if the child is carried out after 8 years).
Age at implantation | 8-10 months,
Age at implantation | 3 years,
Age at implantation | 5 years
Age at implantation | 8 years (or 6 months after surgery if the child is carried out after 8 years).
Distance visual acuity | age of 8 years and 6 months after surgery if the child is carried out after the age of 8.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Robert, MD, Principal Investigator — Hôpital Necker - Enfants Malades, Assistance Publique-Hôpitaux de Paris, France
Locations (1):
- Hospital Necker - Enfants Malades (Assistance Publique-Hôpitaux de Paris), Paris, France